CLINICAL TRIAL: NCT01647607
Title: Young and Strong: An Education and Supportive Care Intervention Study for Young Women With Breast Cancer
Acronym: Y&S
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Dana-Farber Cancer Institute (Other)
Collaborators: American Society of Clinical Oncology (Other)
Responsible Party: Principal Investigator, Ann H. Partridge, MD, MPH, Principal Investigator, Dana-Farber Cancer Institute
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: DFCI 12-101
Record Dates: First submitted 2012-07-19; First posted 2012-07-23 (Estimated); Last update posted 2020-07-29 (Actual); Status verified 2020-07

CONDITIONS: Breast Cancer
Keywords: Breast Cancer; Young Women; Fertility; Physical Activity; Survivorship
MeSH Terms: conditions — Breast Neoplasms; Motor Activity

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Young Women's Intervention (YWI) (Experimental): This arm involves administration of an educational intervention that focuses on issues unique to young women with breast cancer, including career development, starting/raising a family, body image, and genetic predispositions to breast cancer.
  Interventions: Behavioral: Young Women's Intervention (YWI)
- Physical Activity Intervention (PAI) (Active Comparator): This arm involves administration of an educational intervention that focuses on developing and/or maintaining a healthy lifestyle for young women with breast cancer, including the benefits of exercise and resources to enhance physical activity after diagnosis.
  Interventions: Behavioral: Physical Activity Intervention (PAI)

INTERVENTIONS:
Behavioral: Young Women's Intervention (YWI) — This educational intervention uses print and web-based materials to focus on issues unique to young women with breast cancer, including career development, starting/raising a family, body image, and genetic predispositions to breast cancer.
  Arms: Young Women's Intervention (YWI)
Behavioral: Physical Activity Intervention (PAI) — This educational intervention uses print and web-based materials that focus on developing and/or maintaining a healthy lifestyle for young women with breast cancer, including the benefits of exercise and resources to enhance physical activity after diagnosis.
  Arms: Physical Activity Intervention (PAI)

SUMMARY:
The purpose of this study is to address gaps in care of young women with breast cancer by determining whether educational interventions focusing on issues unique to young women with breast cancer and healthy lifestyles for women with breast cancer help to improve care of young breast cancer patients. The investigators believe that if addressed early in a young woman's care, concerns related to fertility, body image, sexual dysfunction, and physical activity will improve the satisfaction with care and quality of life of this vulnerable population. The research will be conducted by exporting refined, previously piloted educational interventions to 14 academic sites and 40 community medical clinics. The investigators will compare how interaction with each intervention affects patients' quality of life and satisfaction with quality of care.

DETAILED DESCRIPTION:
Breast cancer in young women is a not a common disease, yet over 12,000 women under 40 are diagnosed with invasive breast cancer yearly in the United States alone and an additional 2000 are diagnosed with noninvasive disease. Furthermore, when young women are diagnosed with breast cancer, the burden of the disease and treatment on this population is great. Breast cancer is the leading cause of cancer-related deaths in women under 40, and survival rates for young women with breast cancer are lower than for their older counterparts (21,22).

In addition to being at higher risk of dying from breast cancer, and therefore usually receiving more aggressive therapy, young women are at higher risk of distress both at diagnosis and follow-up. Young women with breast cancer face a variety of problems unique to or accentuated by their young age (1). They are more likely to be diagnosed at a stage in life when they fill multiple roles that may not easily be taken over by others (e.g. parenting of young children, completing education, developing a career). Concerns with attractiveness and fertility are often of substantial importance in this population, as many young women are interested in having biologic children following treatment. They also have a greater risk of harboring a genetic risk factor for breast cancer than older patients. Finally, more than older women with breast cancer, who represent the majority of women with the disease, young women often feel isolated and feel that they lack information, and they sometimes are concerned that their doctors are unsure of how to treat them (2,3). Distress may be confounded by a lack of information, provider awareness, peer support, and resources to address young women's concerns, which may contribute to the greater psychosocial distress seen in younger women at both diagnosis and in follow-up compared with older women (4-14). Thus, attention to these concerns in young breast cancer patients is warranted.

Available evidence, however, suggests that attention to important supportive care and survivorship issues including fertility, menopausal concerns, body image, sexual functioning, genetic risk, and psychosocial health have been repeatedly found to be deficient in treatment of young women (15,23-28). Many groups, including ours, have demonstrated that there are substantial inadequacies in attention to fertility and menopausal risks in this population despite recent guidelines recommending their consideration with every young patient (15-20).

Weight gain is another common concern in women diagnosed with breast cancer and has been associated with reductions in physical activity. Studies have demonstrated that 68% of women with early stage breast cancer gain weight after diagnosis and women who receive chemotherapy are at highest risk of weight gain, especially premenopausal women who go through menopause with treatment (33-36). Some evidence suggests that exercise may help prevent treatment-related weight gain and improve psychological outcomes in women diagnosed with early stage breast cancer (38-40). Importantly, exercise and lack of weight gain have been repeatedly associated with improved disease outcomes in breast cancer survivors (41-43).

Again, available evidence suggests the majority of breast cancer survivors do not participate in regular physical activity and that there is clearly room for improvement (43-45). Currently, encouraging physical activity is not a well-recognized standard in breast cancer care, and interventions to assist patients and providers to increase patient exercise behaviors in standard oncology care are needed.

Among older women, access to information and psychosocial support is associated with better quality of life in breast cancer survivors. However, there are no data available to indicate how these processes operate in younger women specifically or what services might mitigate psychosocial distress (29-32). We believe that attention to the issues in young women with breast cancer that are outlined above may be associated with better satisfaction with quality of care and treatment decisions, decreased distress, and better overall quality of life.

To address these critical issues, we have developed a comprehensive Program for Young Women with Breast Cancer at Dana-Farber Cancer Institute (DFCI) to provide additional care, support, and education for young women with breast cancer. Based on the preliminary success of this program, we seek to export this unique model of care to young women with breast cancer who receive care outside of comprehensive cancer centers in an effort to improve the quality of care delivered, the satisfaction with care, and the psychosocial well-being of this vulnerable population.

In the proposed study, we will build on our previous work that developed and piloted an educational and support intervention to improve the quality of care delivered to young women with breast cancer. To achieve these aims, we have created educational interventions focused on issues faced by young women with breast cancer, including but not limited to fertility, satisfaction with care, and physical activity. We will use piloted components of the Program for Young Women with Breast Cancer, as well as piloted exercise intervention materials, to create two educational interventions for this population.

We plan to evaluate both interventions in a randomized controlled trial (RCT) in which community and academic practices and their respective patients will be randomized to an intervention that either focuses on issues unique to young women with breast cancer (Young Women's Intervention, or YWI) or one that focuses on leading a healthy lifestyle as a breast cancer patient (Physical Activity Intervention, or PAI). The rigorous study design of this research will provide important information on the effects of these interventions to improve the care of young women with breast cancer. Therefore, through our intervention, we hope to elucidate what factors might improve quality of life in young women with breast cancer. Ultimately, this work should provide a model for intervening to improve the care of other unique populations.

ELIGIBILITY:
Inclusion Criteria:

* Female age 18-45 years at diagnosis
* Within 3 months of stage I-III invasive breast cancer diagnosis
* No known recurrence of breast cancer or metastatic breast cancer
* Able to read and write in English
* Has first appointment with medical oncologist after the provider's practice is enrolled in the study

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 467 (Actual)
Dates: Start 2012-06; Primary Completion 2015-08 (Actual); Study Completion 2017-12-20 (Actual)

PRIMARY OUTCOMES:
Comparison of attention rates in the YWI and the PAI | 3 Months Post-Enrollment
  The YWI and PAI arms will be compared in terms of the attention rate at 3 months using generalized estimated equations (GEEs) to account for clustered binary data. Comparison will be based on testing the term for treatment arm.

SECONDARY OUTCOMES:
The effect of the YWI on quality of care measures | 3, 6, and 12 Months Post-Enrollment
  To describe the effect of the YWI on other important quality of care measures (attention to genetic issues and attention to emotional health), we will estimate proportions for each arm and report 95% Confidence Intervals (CIs), evaluating the measures separately.
Effect of the PAI on improvement of exercise behaviors | 3 Months Post-Enrollment
  To examine the effects of the PAI on improvement of exercise behaviors, the mean change in MVPA at 3 months (post - pre) will be evaluated in each of the arms. Estimates of mean change and 95% CIs will be determined using GEEs accounting for a stratum effect and clustering within practice.
Effects of the PAI on changes in physical activity based on MVA at three months | 3 Months Post-Enrollment
  To examine the effects of the PAI on change in exercise behaviors based on other measures of physical activity, the mean change in MVA at 3 months and the change in LSI at 3 months will be evaluated in each of the arms. Change at 3 months is change from recalled pre-intervention to 3 months (post - pre). Estimates of mean change and 95% CIs will be determined using GEEs accounting for a stratum effect and clustering within practice.
Relationship between attention rate and quality of care within each arm (YWI and PAI) | 3 Months Post-Enrollment
  To describe the relationship of the attention rate at 3 months with other quality of care measures at 3 months, the quality of care measures will be dichotomized by the median or an established cutoff (high score vs. low score) and the attention rate within each group will be estimated with 95% CIs, accounting for clustering within practice and not for stratification. Quality of care measures will be evaluated separately and relationships will be described for each arm separately.
Effect of demographics on the YWI | 3, 6, and 12 Months Post-Enrollment
  To further describe the YWI treatment effect, exploratory analyses may include adjustment for patient demographics and, if appropriate, including variables in the secondary analyses as well as practice-level characteristics such as setting (urban, suburban, rural) and size of practice.
Effect of the YWI on maintenance of the attention rate | 6 Months Post-Enrollment
  To examine the effects of the YWI on maintenance of the attention rate, we will determine the attention rate at 6 months and 95% CI. There will be separate estimates for each arm.
Effect of the PAI on maintenance of exercise behaviors | 6 and 12 Months Post-Enrollment
  To examine the effects of the PAI on maintenance of exercise behaviors, the arms will be evaluated in terms of mean change in MVPA at 6 and 12 months (post - pre). Time points will be evaluated separately. Descriptive analyses will use GEE models similar to those evaluating change at 3 months.

CONTACTS AND LOCATIONS:
Overall Officials: Ann H Partridge, MD, MPH, Principal Investigator — Dana-Farber Cancer Institute
Locations (4):
- United States (4):
  - University of Colorado, Aurora, Colorado
  - Penrose St. Francis Health Services, Colorado Springs, Colorado
  - Presence Resurrection Medical Center, Chicago, Illinois
  - Albert Einstein Medical Center, Philadelphia, Pennsylvania

REFERENCES:
- [Background] Greaney ML, Sprunck-Harrild K, Ruddy KJ, Ligibel J, Barry WT, Baker E, Meyer M, Emmons KM, Partridge AH. Study protocol for Young & Strong: a cluster randomized design to increase attention to unique issues faced by young women with newly diagnosed breast cancer. BMC Public Health. 2015 Jan 31;15:37. doi: 10.1186/s12889-015-1346-9. PMID 25636332
- [Background] Partridge AH, Ruddy KJ, Barry WT, Greaney ML, Ligibel JA, Sprunck-Harrild KM, Rosenberg SM, Baker EL, Hoverman JR, Emmons KM. A randomized study to improve care for young women with breast cancer at community and academic medical oncology practices in the United States: The Young and Strong study. Cancer. 2019 Jun 1;125(11):1799-1806. doi: 10.1002/cncr.31984. Epub 2019 Feb 1. PMID 30707756
- [Derived] Tesch ME, Sorouri K, Zheng Y, Rosenberg SM, Ruddy KJ, Emmons KM, Dutton MC, Partridge AH. Contraception use and changes in young women with newly diagnosed breast cancer. Fertil Steril. 2025 Mar;123(3):488-498. doi: 10.1016/j.fertnstert.2024.09.024. Epub 2024 Sep 19. PMID 39306190
- [Derived] de Kermadec E, Zheng Y, Rosenberg S, Ruddy KJ, Ligibel JA, Emmons KM, Partridge AH. Fertility concerns and treatment decision-making among national sample of young women with breast cancer. Cancer Med. 2024 Jan;13(1):e6838. doi: 10.1002/cam4.6838. Epub 2023 Dec 22. PMID 38131887
- [Derived] Carroll BR, Zheng Y, Ruddy KJ, Emmons KM, Partridge AH, Rosenberg SM. Satisfaction with Care and Attention to Age-Specific Concerns by Race and Ethnicity in a National Sample of Young Women with Breast Cancer. J Adolesc Young Adult Oncol. 2024 Feb;13(1):105-111. doi: 10.1089/jayao.2023.0068. Epub 2023 Aug 18. PMID 37594766
- [Derived] Cook EE, Rosenberg SM, Ruddy KJ, Barry WT, Greaney M, Ligibel J, Sprunck-Harrild K, Holmes MD, Tamimi RM, Emmons KM, Partridge AH. Prospective evaluation of the impact of stress, anxiety, and depression on household income among young women with early breast cancer from the Young and Strong trial. BMC Public Health. 2020 Oct 6;20(1):1514. doi: 10.1186/s12889-020-09562-z. PMID 33023562